CLINICAL TRIAL: NCT04402515
Title: Preferences and Consequences in Therapy Decision-making: Tiotropium Bromide Plus Olodaterol vs ICS-containing Regimens in COPD Patients in the Portuguese Primary Care Setting: an Observational, Cross-sectional Study
Brief Title: Tiotropium Plus Olodaterol vs Inhaled Corticosteroids (ICS) Regimens in the Portuguese Primary Care Setting (TIOLCOR Study)
Status: Withdrawn | Type: Observational
Why Stopped: not due to safety reasons
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0096
Record Dates: First submitted 2020-05-05; First posted 2020-05-27 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tiotropium plus Olodaterol treatment regimen
  Interventions: Drug: TIO/OLO
- Inhaled corticosteroids-containing treatment regimen
  Interventions: Drug: ICS

INTERVENTIONS:
Drug: TIO/OLO — Tiotropium/Olodaterol
  Groups: Tiotropium plus Olodaterol treatment regimen
Drug: ICS — inhaled cortocosteroids
  Groups: Inhaled corticosteroids-containing treatment regimen

SUMMARY:
What are the differences between patients prescribed a new maintenance treatment for Chronic Obstructive Pulmonary Disease (COPD) with tiotropium/olodaterol (TIO/OLO) or Inhaled Corticosteroids (ICS)-containing regimens in terms of sociodemographic, anthropometric and clinical characteristics?

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 40 years at the date of COPD diagnosis.
2. Diagnosis of COPD confirmed by the investigator. A spirometry confirming the diagnosis (FEV1/forced vital capacity [FVC] ratio <0.7) and performed within the three years prior to the inclusion visit must be available in the patient's medical records.
3. Prescription of a new maintenance COPD treatment with TIO/OLO or ICS-containing regimens (not including TIO/OLO) 3 months (-7/+30 days) prior to the inclusion visit. The COPD treatment may have been prescribed at primary care sites or at the hospital.
4. Written informed consent prior to participation.

Exclusion Criteria:

1. Respiratory disorders other than COPD, such as asthma-COPD overlap or asthma (prior to or at the index date).

2a. For treatment naïve patients (i.e., those who have never started a maintenance therapy for COPD [with either short- or long-acting bronchodilators or ICS]) - no data on the GOLD 2019 group at the index date is available in the medical records. Patients may still be included if the determination of the GOLD 2019 group is possible based on the medical records' data and/or patient interviews (e.g. by using information on exacerbation history in the 12 months prior to the index date, and data on mMRC and COPD Assessment Test (CAT) at the index date).

2b. For treatment experienced patients - no data on the predominant treatable trait to target at the index date (dyspnea, exacerbation or both) is available in the medical records. Patients may still be included if this information is obtained based on patient interviews.

3. Participation in a clinical trial within the 3 months prior to the inclusion visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population are COPD patients starting a new maintenance COPD treatment with TIO/OLO or with an ICS-containing regimen in the primary care setting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-28 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
N of patients by education level | up to 4 months
smoking status | up to 4 months
BMI | up to 4 months
N of patients by Portugal region | up to 4 months
  regions: North, Center, Lisbon, Alentejo and Algarve (NUTS II)
year of COPD diagnosis | up to 4 months
comorbidities | up to 4 months
GOLD 2019 group assessment | up to 4 months
  Global Initiative for Chronic Obstructive Lung Disease; groups A, B, C, D
GOLD 2019 grade | up to 4 months
  Global Initiative for Chronic Obstructive Lung Disease; grades 1-4
blood eosinophil count | up to 4 months
post-bronchodilator FEV1/FVC ratio (FEV1/FVC) ratio | up to 4 months
  FEV1: Forced expiratory volume in one second; FVC: Forced Vital Capacity
FEV1 % predicted | up to 4 months
number of COPD exacerbations | in the 12 months prior to the index date
N of patients with pneumonia | up to 4 months
Patient symptomatology according to the modified British Medical Research Council (mMRC) questionnaire | up to 4 months
CAT score | up to 4 months
  CAT: COPD Assessment Test
Setting in which the COPD treatment was prescribed | up to 4 months
  primary vs. hospital
Reasons for COPD treatment change | Index date
  Index date is the prescription date of the new or initial COPD maintenance treatment.
Reasons for COPD treatment change between the index date and the inclusion visit | up to 4 months

SECONDARY OUTCOMES:
Number of patients for whom the new COPD treatment is in accordance with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 Guideline recommendations | Index date
  Index date is the prescription date of the new or initial COPD maintenance treatment.
Patient Quality of Life according to EQ-5D-5L questionnaire | up to 4 months
Overall patient satisfaction with inhaler device according to a 5-point Likert scale | up to 4 months
Patient satisfaction with treatment according to Treatment Satisfaction Questionnaire for Medication | up to 4 months

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com